CLINICAL TRIAL: NCT05819840
Title: Vascular Structure, Vascular Function and Vascular Aging in Adults Diagnosed With Persistent COVID. ICOPER Study.
Brief Title: Vascular Structure, Vascular Function and Vascular Aging in Adults Diagnosed With Persistent COVID
Acronym: ICOPER
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fundacion para la Investigacion y Formacion en Ciencias de la Salud (Other)
Responsible Party: Sponsor
Other Study IDs: GRS2501/B/22
Record Dates: First submitted 2023-04-18; First posted 2023-04-19 (Actual); Last update posted 2023-06-29 (Actual); Status verified 2023-04

CONDITIONS: Persistent COVID-19; Quality of Life; Lifestyles; Arterial Stiffness
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — The analytical data closest to the patient's clinical history prior to SARS-CoV-2 infection will be collected, and the analytical data during the acute SARS-CoV-2 infection, including basal glycemia, HbA1c, TSH, profile lipid, complete blood count, liver profile, creatinine and creatinine albumin index, Vit D and PCR. At the time of inclusion, a fasting test will be carried out, including basal glycemia, HbA1c, TSH, lipid profile, complete blood count, liver profile, creatinine and creatinine albumin index, Vit D, ESR, CRP and interleukins.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The ICOPER study aims to analyze the structure, vascular function, vascular aging and determining factors in 300 adults diagnosed with Persistent Covid in the field of Primary Health Care.

DETAILED DESCRIPTION:
Objective: To analyze the structure, the vascular function, the vascular aging and the determining factors in adults with a diagnosis of Persistent Covid and the differences by gender.

Design: Cross-sectional descriptive observational study. Setting: The study will be carried out at the Salamanca Primary Care Research Unit (APISAL). Study Subjects: The study includes the basis of the Persistent Covid Monographic consultation in the Internal Medicine Service of the University Hospital of Salamanca and the subjects with the diagnosis of Persistent Covid in the MEDORA Primary Care clinical history. Thus, 300 subjects have been obtained who are diagnosed with Persistent Covid, who meet the diagnostic criteria established by the Spanish Society of General and Family Physicians and sign the informed consent.

Measurements: The variables reflected in the Integrated Assistance process for the Care of People Affected by SARS CoV-2 of the Junta de Castilla y León will be collected, to evaluate the functional status of the patient and persistent symptoms, their impact on activities of daily life and quality of life of patients with Persistent Covid and the perception of their health. Lifestyles (diet, physical activity, tobacco and alcohol), psychological factors and cognitive impairment will be collected using validated questionnaires, and physical activity will be objectively measured with a 7-day pedometer. Vascular structure and function will be analyzed by measuring the thickness of the carotid intima media (Sonosite Micromax); pulse wave analysis and carotid-femoral pulse wave velocity (VOPcf) (Sphygmocor System). Cardio Ankle Vascular Index (CAVI), ankle-brachial pulse wave velocity (VOPbt) and ankle-brachial index (Vasera VS-2000®). Vascular aging will be calculated using the 10 and 90 percentiles of the VOPcf and the VOPbt. Demographic, analytical variables and to assess retinal, cardiac, renal, cerebral vascular lesion and cardiovascular risk will be collected.

ELIGIBILITY:
Inclusion Criteria:

* History of probable or confirmed SARS-CoV-2 infection, usually 3 months after onset, with symptoms that last at least 2 months and cannot be explained by an alternative diagnosis.
* Common symptoms should include fatigue, shortness of breath, and cognitive dysfunction, and an impact on daily functioning.

Exclusion Criteria:

* Subjects in a terminal situation.
* Inability to travel to health centers.
* Presenting a history of cardiovascular disease (ischemic heart disease or cerebrovascular disease).
* Glomerular filtration rate of less than 30%.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Through consecutive sampling, 300 subjects will be selected who meet the WHO clinical definition of Persistent Covid established by international Delphi consensus. The subjects will be recruited from the existing records in the Primary Care consultations and in the Internal Medicine Persistent Covid consultation in the Salamanca health area.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-03-09 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Pulse Wave Velocity | 1 year
  Measurement by SphygmoCor System (meters/seg)

SECONDARY OUTCOMES:
Carotid intima-media thickness (IMT) | 1 year
  Measurement by Sonosite Micromax Ultrasound (mm)
Cardio Ankle Vascular Index (CAVI) | 1 year
  Measurement by Vasera device 2000 (not units)
Physical Activity | 1 year
  World Questionnaire on Physical Activity (GPAQ)
Eating habits | 1 year
  Mediterranean Diet Adherence PREDIMED Questionnaire
Smoking | 1 year
  Measurement by a questionnaire of four questions adapted from the WHO MONICA study
Drinking habits | 1 year
  Measurement by a frequency alcohol questionnaire (units/day)
Psychological factors | 1 year
  Goldberg Anxiety and Depression Scale
Cognitive evaluation | 1 year
  Measurement by Montreal Cognitive Assessment (MOCA) (points). Range: 0-30 points. A score of 26 points or above is considered normal.

CONTACTS AND LOCATIONS:
Locations (1):
- Primary Care Research Unit of Salamanca (APISAL), Salamanca, Spain

REFERENCES:
- [Derived] Vicente-Gabriel S, Lugones-Sanchez C, Tamayo-Morales O, Vicente Prieto A, Gonzalez-Sanchez S, Conde Martin S, Gomez-Sanchez M, Rodriguez-Sanchez E, Garcia-Ortiz L, Gomez-Sanchez L, Gomez-Marcos MA; EVA-Adic Investigators Group. Relationship between addictions and obesity, physical activity and vascular aging in young adults (EVA-Adic study): a research protocol of a cross-sectional study. Front Public Health. 2024 Jan 26;12:1322437. doi: 10.3389/fpubh.2024.1322437. eCollection 2024. PMID 38344236
- [Derived] Gomez-Sanchez L, Tamayo-Morales O, Suarez-Moreno N, Bermejo-Martin JF, Dominguez-Martin A, Martin-Oterino JA, Martin-Gonzalez JI, Gonzalez-Calle D, Garcia-Garcia A, Lugones-Sanchez C, Gonzalez-Sanchez S, Jimenez-Gomez R, Garcia-Ortiz L, Gomez-Marcos MA, Navarro-Matias E; ICOPER investigators group. Relationship between the structure, function and endothelial damage, and vascular ageing and the biopsychological situation in adults diagnosed with persistent COVID (BioICOPER study). A research protocol of a cross-sectional study. Front Physiol. 2023 Sep 12;14:1236430. doi: 10.3389/fphys.2023.1236430. eCollection 2023. PMID 37772064